CLINICAL TRIAL: NCT00568425
Title: Quality of Life and Functional Outcomes After Combined Modality Therapy for Anal Cancer: A Comparison of Conventional Versus Intensity-Modulated Radiation Therapy (ANAL0002)
Brief Title: QOL & Functional Outcomes After Combined Modality Tx for Anal CA: Comparison of Conventional vs IMRT
Status: Terminated | Type: Observational
Why Stopped: Inadequate response to Scientific Review Committee.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-03103; 96405 (Other: Stanford University Alternate IRB Approval Number); SU-11062007-812 (Other: Stanford University); ANAL0002 (Other: OnCore); NCT00533325 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is show that intensity-modulated radiotherapy (IMRT), as compared with conventional radiotherapy, improves the precision of tumor targeting and reduces the acute and late effects of radiation toxicity when used to treat anal cancer. Results from this work will provide a basis for incorporating the use of IMRT to treat anal cancer in future treatment protocols.

DETAILED DESCRIPTION:
The objectives of this study are three-fold. First, we would like to learn and compare the doses of radiation received by the tumor and the normal tissues in anal cancer patients treated with IMRT, and in those treated with conventional radiotherapy. Second, we wish to compare the acute effects of radiation treatment in both groups of patients. Our third objective is to evaluate the late effects of radiation treatment in both groups of patients. The first two objectives will be studied using a retrospective analysis of patients with anal cancer treated at Stanford University Medical Center. The third objective will require these patients to complete and return three quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:Histologically confirmed diagnosis of squamous cell carcinoma of the anus. Must be able to provide informed consent. Exclusion Criteria:History of new malignancy since the time of treatment for anal cancer. Non-English speaking.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed diagnosis of squamous cell carcinoma of the anus
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the late effects of radiation treatment | one day
  Quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lane Welton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States